CLINICAL TRIAL: NCT00047125
Title: Randomized Phase III Study On The Selection Of The Target Volume In Postoperative Radiotherapy For Cervical Lymph Node Metastases Of Squamous Cell Carcinoma From And Unknown Primary (CUP)
Brief Title: Radiation Therapy in Treating Patients With Metastases to the Lymph Nodes in the Neck From an Unknown Primary Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Radiation Therapy Oncology Group (Network); NCIC Clinical Trials Group (Network); Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-24001-22005; EORTC-24001; EORTC-22005; DAHANCA-EORTC-24001; CAN-NCIC-EORTC-24001; RTOG-EORTC-24001
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma of Unknown Primary
Keywords: newly diagnosed carcinoma of unknown primary; squamous cell carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective irradiation (Experimental): Irradiation of the ipsilateral level I - V of the neck up to a dose of 60 Gy (30x2Gy in 6 weeks).
  Interventions: Radiation: radiation therapy
- Extensive irradiation + ipsilaterals levels (Active Comparator): Irradiation on the whole mucosa of the larynx, hypopharynx, oropharynx and nasopharynx, and on both sides of the neck (levels I -V) up to a prophylactic dose of 50 Gy (25 x 2 Gy in 5 week).Irradiation of the ipsilateral level I - V of the neck should continue with an additional 10 Gy boost for a total dose of 60 Gy (30 x 2 Gy in 6 weeks).
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy in different ways may kill more tumor cells. It is not yet known which regimen of radiation therapy is more effective in treating patients who have metastases to the lymph nodes in the neck.

PURPOSE: Randomized phase III trial to compare different radiation therapy regimens in treating patients who have metastases to the lymph nodes in the neck from an unknown primary tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival of patients with cervical lymph node metastases of squamous cell carcinoma from an unknown primary treated with selective irradiation vs extensive irradiation.
* Compare the overall survival of patients treated with these regimens.
* Compare the incidence of acute and late side effects in the head and neck region in patients treated with these regimens.
* Compare control of the neck and incidence of subsequent primary in the head and neck region in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to disease stage (N1-2a vs N2b-3), radiation technique (2D vs 3D conformal vs intensity-modulated), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo selective irradiation of the ipsilateral level of the neck once daily 5 days a week for 6 weeks.
* Arm II: Patients undergo extensive irradiation of the neck (nasopharyngeal, oropharyngeal, hypopharyngeal, and laryngeal mucosa and ipsilateral neck node areas on both sides of the neck) once daily 5 days a week for 6 weeks.

In both arms, treatment continues in the absence of unacceptable toxicity or disease progression.

Quality of life is assessed at baseline, at week 4, on the last day of therapy, and then every 3 months for 1 year.

Patients are followed at day 30, every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 600 patients (300 per treatment arm) will be accrued for this study within 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma in cervical lymph node metastasis from an unknown primary tumor

  * Histopathological grade WHO 1-3
  * Pathological stage N1, N2a, N2b, or N3
  * No N2c (i.e., bilateral metastatic nodes)
  * No single node in supraclavicular fossa or submandibular area
  * No evidence of primary tumor in head and neck, lung, esophageal, or other site
* Prior radical, radical modified, or extended radical dissection within the past 8 weeks

  * Selective neck dissection allowed (surgeon must justify why standard procedure was not performed)
  * No node excision alone
  * R0 or R1 disease after dissection
* No distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able and willing to complete quality of life questionnaires
* No other prior or concurrent malignancy except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Concurrent chemotherapy allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No other prior therapy for carcinoma of unknown primary except neck dissection

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2002-07; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Vincent G. Gregoire, MD, PhD, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Sharon A. Spencer, MD, Study Chair — University of Alabama at Birmingham; Samy El-Sayed, MD, FFR, FRCR, FRCP, Study Chair — Ottawa Regional Cancer Centre; Esat M. Ozsahin, MD, PhD, Study Chair — Centre Hospitalier Universitaire Vaudois; Cai Grau, MD, Study Chair — Aarhus Universitetshospital - Aarhus Sygehus
Locations (262):
- United States (237):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Montgomery Cancer Center, Montgomery, Alabama
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiation Oncology Centers - Sacramento, Sacramento, California
  - Radiation Medical Group, Incorporated, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - St. Joseph's Regional Cancer Center, Stockton, California
  - Torrance Memorial Medical Center, Torrance, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Hospital of St. Raphael, New Haven, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Florida Radiation Oncology Group, Jacksonville, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - CCOP - Scott and White Hospital, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Cancer Center at St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Cancer Center at Lexington Clinic, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Louisville Radiation Oncology Center at Caritas Regional Cancer Center, Louisville, Kentucky
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - NSMC Cancer Center, Peabody, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Medical Center of Princeton, Princeton, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Lourdes Regional Cancer Center, Binghamton, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - North Shore Radiation Oncology, Setauket, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Cancer Center at Christ Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Frank C. Love Cancer Institute at St. Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Dale and Frances Hughes Cancer Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes-Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Arlington Cancer Center, Arlington, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Cancer Institute at Virginia Mason Medical Center, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Clinique Sainte Elisabeth, Namur
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre at Regional Hospital of Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Care, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Aarhus University Hospital - Aarhus Sygehus, Aarhus, Denmark
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland